CLINICAL TRIAL: NCT03178799
Title: Fracture Liaison Service：A Randomized Control Trial
Brief Title: Randomized Fracture Liaison Services
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201703023RINC
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis Fracture
Keywords: Fractures; Osteoporosis; Care management; cost-effeciveness; Randomized controlled trial
MeSH Terms: conditions — Osteoporotic Fractures; Fractures, Bone; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FLS: Fracture Liaison Service (Care managers based coordination service for fragility fracture patients with followed up telephone call at 4, 8, 12, 18, 24 months then annually for up to 10 years (to 2028).)
- UC: usual care (Care managers will perform baseline assessments and follow them by telephone annually for up to 10 years (to 2028). )

SUMMARY:
Aims: To compare clinical outcomes for patients under FLS and usual care at the NTUH MH and BB.

Method: Four hundred subjects with new hip fracture or newly identified vertebral fracture are randomly assigned into FLS and usual care (UC). FLS subjects received osteoporosis-related assessments, treatments, consultations on diet, medications, exercise, fall preventions given mainly by care managers with followed up telephone call at 4, 8, 12, 18, 24 months then annually for up to 10 years. Care managers will perform baseline assessments and follow them by telephone annually for up to 10 years for UC subjects. Major outcomes include bone mineral density assessment rate, calcium, vitamin D, and osteoporosis medication initiation and adherence rate, fall and fracture incidences, mortality, and healthcare resource utilizations.

DETAILED DESCRIPTION:
Background: First fragility fracture increased risk for further fracture for 2-4 folds. However, most fracture sufferers did not receive secondary prevention for osteoporosis to decrease future fracture risks. Since 2014, the National Taiwan University Hospital (NTUH) Healthcare system established fracture liaison services and were certified as gold (main hospital, MH) and silver (Beihu branch, BB) medal for best practices. Our preliminary results showed that compared with national average data, hip fracture patients under FLS may have lower mortality rate. However, randomized control trial (RCT) is still needed to confirm results from observational studies.

Aims: to compare clinical outcomes for patients under FLS and usual care at the NTUH MH and BB.

Method: Four hundred subjects with new hip fracture or newly identified vertebral fracture are randomly assigned into FLS and usual care (UC). FLS subjects received osteoporosis-related assessments, treatments, consultations on diet, medications, exercise, fall preventions given mainly by care managers with followed up telephone call at 4, 8, 12, 18, 24 months then annually for up to 10 years. Care managers will perform baseline assessments and follow them by telephone annually for up to 10 years for UC subjects. Major outcomes include bone mineral density assessment rate, calcium, vitamin D, and osteoporosis medication initiation and adherence rate, fall and fracture incidences, mortality, and healthcare resource utilizations.

Anticipated results: Provide evidence on benefit of FLS in RCT on osteoporosis evaluation, medication initiation, mediation adherence, calcium, vitamin D, protein, exercise adherence, fall, re-fracture, mortality and other outcomes.

ELIGIBILITY:
Inclusion criteria：

* Age>=50
* New hip fracture from orthopedic ward
* Newly identified vertebral fracture (either morphological or clinical)/ old hip fracture without osteoporosis treatment referred by team physicians either inpatients or outpatients
* Willing to accept 10 years of follow-ups.

Exclusion criteria

* Traumatic or pathologic fractures
* Atypical femoral shaft fracture
* Participating in other medication intervention trials
* Less than 2 years of life expectancy judged by team physicians
* Incapable of accepting evaluation for cognitive, communication, and physical problems judged by team physicians or coordinators.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four hundred subjects with new hip fracture or newly identified vertebral fracture are randomly assigned into FLS and usual care (UC). FLS subjects received osteoporosis-related assessments, treatments, consultations on diet, medications, exercise, fall preventions given mainly by care managers with followed up telephone call at 4, 8, 12, 18, 24 months then annually for up to 10 years. Care managers will perform baseline assessments and follow them by telephone annually for up to 10 years for UC subjects.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis Medication Adherence Rate at 24 months | 24 months
  Defined at percents of osteoporosis medication use/expected osteoporosis medication prescriptions in 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided